CLINICAL TRIAL: NCT00380146
Title: An Open-label in Vivo Drug Study to Evaluate the Pharmacokinetics, Therapeutic Efficacy, Gametocyte Carriage and Birth Outcomes Following Sulfadoxine-pyrimethamine Intermittent Presumptive Treatment (SP IPT) in Pregnant Women
Brief Title: Pharmacokinetics, Efficacy, Gametocyte Carriage, Birth Outcomes Following Sulfadoxine-pyrimethamine Intermittent Presumptive Treatment in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Karen I Barnes (Other)
Collaborators: Global Fund (Other); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor-Investigator, Professor Karen I Barnes, Professor, Clinical Pharmacology, University of Cape Town
Organization: University of Cape Town (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SEACAT2.2
Record Dates: First submitted 2006-09-22; First posted 2006-09-25 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Malaria
Keywords: Malaria; Intermittent presumptive treatment; IPT; Pharmacokinetic; Efficacy; Gametocyte; Molecular markers
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SP plus artesunate (Experimental): SP (Fansidar®, Roche South Africa) at a dose of 25/1.25mg/kg of sulfadoxine/pyrimethamine respectively on day 0 only, and artesunate (Arsumax®, Sanofi-Aventis, South Africa) at a dose of 4mg/kg on days 0, 1, and 2
  Interventions: Drug: sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine

SUMMARY:
The main purpose of this study is to compare the drug levels of sulfadoxine-pyrimethamine found when given to pregnant women for the prevention of malaria to those found in pregnant women given the same drug with artesunate for the treatment of malaria, and also with those drug levels found in non-pregnant women in other malaria treatment studies.

DETAILED DESCRIPTION:
Pregnancy increases the risk of malaria progression and complications with up to a 10-fold increase in the malaria case fatality rate in areas of low transmission. Sulfadoxine-pyrimethamine (SP) is used widely in Africa for the systematic intermittent presumptive, or preventive, treatment (IPTp) during the second and third trimester of pregnancy and a national program of IPTp with SP has been implemented recently in Mozambique. There is evidence that the kinetics of several other antimalarial drugs are altered in pregnancy to the extent that doses are not adequate in pregnancy, however no published study has included a pharmacokinetic component to confirm that standard doses of SP are optimal in this vulnerable patient group. This study therefore creates the opportunity to study whether the pharmacokinetic properties of SP are altered by physiological changes that occur during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female, older than 18 years, > 35kg.
* Gestational age > 16 weeks (fundal height > 16cm) and below 36 weeks gestation.
* Documented informed consent.
* Lives close enough to the study site for reliable follow up and is willing to attend ANC and follow-up visits regularly.

Exclusion Criteria:

* Diagnoses of uncomplicated acute P. falciparum malaria parasitaemia
* Has received anti-malarial treatment in the past 7 days and/or sulfadoxine-pyrimethamine in the past 28 days.
* Known hepatic or renal impairment
* Has received chloramphenicol, cotrimoxazole or tetracyclines (including doxycycline) in the past 7 days or is likely to require these during the study period.
* History of G6PD deficiency.
* Has a history of allergy to any of the study drugs (including other sulphonamides e.g. cotrimoxazole).
* Serious underlying disease that in the opinion of the clinic team and/or Principal Investigator would make the patient unsuitable for the study in terms of their safety or study analysis.
* Imminent delivery expected.
* Prior inclusion in this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-09; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters by measurement of whole blood levels of sulfadoxine and pyrimethamine and plasma levels of artesunate to determine Cmax, Tmax, AUC, half life, volume of distribution and clearance | 0 hours (pre treatment) and repeated on day 0 or 1 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours, and days 2, 3, 7, 14, 21, 28 and 42

SECONDARY OUTCOMES:
Correlation of treatment outcome and gametocyte carriage with pharmacokinetic parameters and pregnancy status | 0 hours (pre treatment) and repeated on day 0 or 1 at 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 hours, and days 2, 3, 7, 14, 21, 28 and 42 , and time of birth outcome
Correlation of frequency of DHFR mutations at codons 436, 437, 540 and 581 in maternal and placental samples with treatment outcomes | Day 42 (or day of withdrawal)
Birth outcomes in terms of major congenital abnormalities, spontaneous abortions, still births and neonatal deaths, gestational age and birth weight, placental weight, newborn head circumference, arm circumference and neurological development | Day of birth outcome
Risk of harm by describing all adverse events and their causality assessments and changes in full blood count, glucose, bilirubin, creatinine, urea and ALT | Days 3, 7, 14, 21, 28 and every 2 weeks thereafter until birth (for a minimum of 42 days) or withdrawal visit
Capacity building by describing the training and development of study teams and their subsequent skills attained | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Karen I Barnes, MBChB, Principal Investigator — University of Cape Town
Locations (1):
- Ndlavela Health Centre, Ndlavela, Maputo, Mozambique